CLINICAL TRIAL: NCT05472948
Title: Surufatinib and Sintilimab in Combination With Capecitabine for Previously Treated Metastatic Small Bowel Adenocarcinoma and Appendiceal Carcinoma: A Single-arm, Multi-center, Phase Ib/II Trial
Brief Title: Surufatinib and Sintilimab in Combination With Capecitabine for Metastatic Adenocarcinoma of Small Intestine or Appendix Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Director of Medical Oncology, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-23
Record Dates: First submitted 2022-07-22; First posted 2022-07-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-06

CONDITIONS: Adenocarcinoma of Small Intestine; Appendix Carcinoma; Metastatic
MeSH Terms: conditions — Appendiceal Neoplasms; Neoplasm Metastasis | interventions — surufatinib; sintilimab; Capecitabine

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib and Sintilimab in Combination With Capecitabine (Experimental): Patients were given solventinib (a "3+3" design was adopted in the dose exploration phase, with two dose levels of 200mg and 250mg for dose exploration; after the recommended dose was determined in the dose exploration phase, the dose amplification phase was entered), once a day (QD) for continuous administration
  * sindilizumab, 200mg, iv every 3 weeks (Q3W)
  * Capecitabine, 1000mg/m2, twice a day (BID, once in the morning and once in the evening), orally after meals, stopped for 1 week after 2 weeks of treatment;
  The three-drug combination therapy was continued every 3 weeks in a cycle until patients developed disease progression or met other criteria for termination of study treatment specified in the protocol.
  Interventions: Drug: Surufatinib; Drug: Sintilimab; Drug: Capecitabine

INTERVENTIONS:
Drug: Surufatinib — Surufatinib will be given 200/250 mg po. qd.
  Other Names: SULANDA
Drug: Sintilimab — Sintilimab administered IV at a dose of 200mg every 3 weeks.
  Other Names: IBI308
Drug: Capecitabine — Capecitabine will be given 2 weeks on/1 week off (1000 mg/m2 BID po.)
  Other Names: Capecitabine tablets

SUMMARY:
To explore the safety and efficacy of Surufatinib and Sintilimab in Combination With Capecitabine in Patients With Previously Treated Metastatic Adenocarcinoma of Small Intestine or Appendix Carcinoma : a Single-arm, a Single-center , Phase 2 Trial. Meanwhile, Exploring the maximum tolerant dose or recommended II research dose of Surufatinib combined with a fixed dose of Sintilimab and Capecitabine using 3 + 3 dose climbing experiment.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological documentation of adenocarcinoma of Small Intestine or Appendix Carcinoma. All other histological types are excluded.
2. Subjects with metastatic adenocarcinoma of Small Intestine or Appendix Carcinoma.
3. Subjects must have failed at least one line of prior treatment.
4. Progression during or within 3 months following the last administration of approved standard therapies . 4.1 Subjects an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy. 4.2 Subjects who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of treatment and precluding retreatment with the same agent prior to progression of disease will also be allowed into the study. 4.3 Subjects may have received prior treatment with Avastin (bevacizumab)
5. Subjects must have measurable or non measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 1.
7. Life expectancy of at least 3 months.
8. Adequate bone marrow, liver and renal function as assessed by the laboratory required by protocol.

Exclusion Criteria:

1. Prior treatment with Surufatinib
2. Previously received anti-programmed death-1 (PD-1) or its ligand (PD-L1) antibody, anti-cytotoxic T lymphocyte-associated antigen 4 (cytotoxic T- lymphocyte-associated Protein 4, CTLA-4) antibody or other drug/antibody that acts on T cell costimulation or checkpoint pathways.
3. Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
4. Cardiological disease including Congestive heart failure, Unstable angina, Myocardial infarction, Cardiac arrhythmias requiring anti-arrhythmic therapy.
5. Uncontrolled hypertension. (Systolic blood pressure 150 mmHg or diastolic pressure 90 mmHg despite optimal medical management).
6. Pleural effusion or ascites that causes respiratory compromise. Arterial or venous thrombotic or embolic events.
7. Any history of or currently known brain metastases.
8. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
9. Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 4 week.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 year
  The PFS is defined as the time from the start of treatment to the date of first documented PD or death as a result of any cause, whichever occurred first. When a patient was alive and without progression, PFS was censored at the date of the last disease assessment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 year
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR).
Overall Survival (OS) | 2 year
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Disease Control Rate (DCR) | 2 year
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD); CR, PR, or SD had to be maintained for at least 28 days from the first demonstration of that rating)
Safety variables (Incidence of Adverse Events [Safety and Tolerability]) | 2 year
  Safety variables will be summarized using descriptive statistics based on adverse events collection

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, Ph.D, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No